CLINICAL TRIAL: NCT05310084
Title: A PHASE 3, RANDOMIZED, OBSERVER-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF BNT162b2 WHEN COADMINISTERED WITH SEASONAL INACTIVATED INFLUENZA VACCINE (SIIV) IN ADULTS 18 THROUGH 64 YEARS OF AGE
Brief Title: Safety and Immunogenicity of BNT162b2 Coadministered With SIIV in Adults 18 Through 64 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4591030; NCT06137001 (obsolete NCT alias)
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an Observer-Blind Study. The vaccines and placebo will be administered by an unblinded third-party site staff member.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Coadministration Group (Experimental): BNT162b2 and SIIV followed by placebo a month later
  Interventions: Biological: BNT162b2; Other: Placebo; Biological: Seasonal Inactivated Influenza Vaccine
- Separate Administration Group (Experimental): Placebo and SIIV followed by BNT162b2 a month later
  Interventions: Biological: BNT162b2; Other: Placebo; Biological: Seasonal Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular injection
Other: Placebo — Saline intramuscular injection
Biological: Seasonal Inactivated Influenza Vaccine — SIIV intramuscular injection

SUMMARY:
This study will assess the safety and immunogenicity of a fourth dose (booster) of BNT162b2 when coadministered with SIIV compared to separate administration of the vaccines when given 1 month apart (SIIV followed by BNT162b2), in participants who have received 3 prior doses of 30 µg BNT162b2, with the third dose being at least 90 days before Visit 1 (Day 1).

* Healthy adults 18 through 64 years of age will be randomized 1:1 to either the co-administration group, or the separate administration group
* The duration of the study for each participant will be approximately 2 months
* There are 3 scheduled study visits each about 1 month apart
* The study will be conducted in New Zealand and Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 18 through 64 years of age, inclusive, at the time of consent.
2. Are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Adults determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study, including adults with preexisting stable disease, defined as disease not requiring significant change in therapy in the previous 6 weeks or hospitalization for worsening disease within 12 weeks before receipt of study intervention.
4. Have received 3 prior doses of 30 µg BNT162b2, with the third dose being at least 90 days before Visit 1 (Day 1). Documented confirmation of prior BNT162b2 receipt must be obtained prior to randomization.
5. Capable of giving personal signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Other medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
2. Allergy to egg proteins (egg or egg products) or chicken proteins.
3. History of Guillain-Barré syndrome.
4. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
5. A positive SARS-CoV-2 test result (either by NAAT or rapid antigen test) within 28 days of Visit 1 (Day 1).
6. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
7. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
8. Women who are pregnant or breastfeeding.
9. Vaccination with any influenza vaccine <6 months before study intervention administration, or planned receipt of any licensed or investigational nonstudy influenza vaccine during study participation.
10. Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), eg, for COPD, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
11. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
12. Receipt of any passive antibody therapy specific to COVID-19 from 90 days before study intervention administration or planned receipt throughout the study.
13. Prior receipt of any COVID-19 vaccine other than BNT162b2 or receipt of more than 3 prior doses of BNT162b2.
14. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
15. Investigator site staff or Pfizer/BioNTech employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1134 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- Australia (7):
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Australian Clinical Research Network, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Paratus Clinical Research Brisbane, Albion, Queensland
  - AusTrials - Wellers Hill, Wellers Hill, Queensland
  - Emeritus Research, Camberwell, Victoria
  - Barwon Health, Geelong, Victoria
- New Zealand (19):
  - New Zealand Clinical Research (Auckland), Grafton, Auckland
  - Optimal Clinical Trials, Grafton, Auckland
  - Southern Clinical Trials Totara, New Lynn, Auckland
  - Lakeland Clinical Trials Culloden, Papamoa Beach, Bay of Plenty
  - Pacific Clinical Research Network - Rotorua, Rotorua, Bay of Plenty
  - P3 Research - Tauranga, Tauranga, Bay of Plenty
  - New Zealand Clinical Research (Christchurch), Christchurch, Canterbury
  - Pacific Clinical Research Network - Forte, Christchurch, Canterbury
  - P3 Research - Hawke's Bay, Havelock North, Hawke's Bay Region
  - P3 Research - Palmerston North, Palmerston North, Manawatu-Wanganui
  - Lakeland Clinical Trials Waikato, Hamilton, Waikato Region
  - Lakeland Clinical Trials Wellington, Ebdentown. Upper Hutt, Wellington Region
  - P3 Research - Kapiti, Paraparaumu, Wellington Region
  - Southern Clinical Trials Waitemata Ltd, Auckland
  - Aotearoa Clinical Trials, Auckland
  - Middlemore Clinical Trials, Auckland
  - Southern Clinical Trials Tasman, Nelson
  - Capital, Coast and Hutt Valley District - Wellington Regional Hospital, Wellington
  - P3 Research - Wellington, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murdoch L, Quan K, Baber JA, Ho AWY, Zhang Y, Xu X, Lu C, Cooper D, Koury K, Lockhart SP, Anderson AS, Tureci O, Sahin U, Swanson KA, Gruber WC, Kitchin N; C4591030 Clinical Trial Group. Safety and Immunogenicity of the BNT162b2 Vaccine Coadministered with Seasonal Inactivated Influenza Vaccine in Adults. Infect Dis Ther. 2023 Sep;12(9):2241-2258. doi: 10.1007/s40121-023-00863-5. Epub 2023 Sep 12. PMID 37698774
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1165 participants were screened, out of which 31 were screen failures and 1134 were randomized into the study.
Groups:
- Coadministration Group: Participants were randomized to receive 30 mcg IM injection of BNT162b2 vaccine along with IM injection of SIIV on Day 1 (Visit 1), and IM injection of Placebo 1 month later (Visit 2).
- Separate Administration Group: Participants were randomized to receive an IM injection of Placebo along with IM injection of SIIV on Day 1 (Visit 1), and 30 mcg IM injection of BNT162b2 vaccine 1 month later (Visit 2).
Period: Overall Study
Arm/Group | Coadministration Group | Separate Administration Group
Started | 568 | 566
Vaccinated | 564 | 564
Completed | 560 | 555
Not Completed | 8 | 11
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Participant availability | 0 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Randomized but not vaccinated | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any of the study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Coadministration Group | Separate Administration Group | Total
Number analyzed (Participants) | 564 | 564 | 1128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.7 (13.20) | 39.8 (13.52) | 39.7 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 356 | 361 | 717
  Male | 208 | 203 | 411
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 539 | 537 | 1076
  Unknown or Not Reported | 20 | 18 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 73 | 66 | 139
  Native Hawaiian or Other Pacific Islander | 26 | 36 | 62
  Black or African American | 1 | 2 | 3
  White | 446 | 439 | 885
  More than one race | 1 | 10 | 11
  Unknown or Not Reported | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions included redness, swelling, and pain at the injection site occurring at the BNT162b2 or placebo injection site. Local reactions were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: greater than (>) 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, severe: >10.0 cm, and potentially life threatening (Grade 4): necrosis or exfoliative dermatitis. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity, and potentially life threatening (Grade 4): emergency room visit or hospitalization for severe pain. Exact 2-sided confidence interval (CI), based on the Clopper and Pearson method was used.
Time Frame: Within 7 Days After Vaccination 1
Population: Safety population included all participants who received any of the study intervention. Here, ''Number of participants analyzed'' (N) signifies number of participants evaluable and "Number Analyzed" (n) signifies number of participants evaluable for specified rows for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Coadministration Group: Participants were randomized to receive 30 microgram (mcg) intramuscular (IM) injection of BNT162b2 vaccine along with IM injection of Seasonal Inactivated Influenza Vaccine (SIIV) on Day 1 (Visit 1), and IM injection of Placebo 1 month later (Visit 2).
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 564 | 563
Percentage of participants
  Redness: Any: number analyzed (Participants) | 564 | 562
  Redness: Any | 7.6 [5.6 to 10.1] | 0.5 [0.1 to 1.6]
  Redness: Mild: number analyzed (Participants) | 564 | 562
  Redness: Mild | 6.2 [4.4 to 8.5] | 0.5 [0.1 to 1.6]
  Redness: Moderate: number analyzed (Participants) | 564 | 562
  Redness: Moderate | 1.2 [0.5 to 2.5] | 0 [0.0 to 0.7]
  Redness: Severe: number analyzed (Participants) | 564 | 562
  Redness: Severe | 0.2 [0.0 to 1.0] | 0 [0.0 to 0.7]
  Redness: Grade 4: number analyzed (Participants) | 564 | 562
  Redness: Grade 4 | 0 [0.0 to 0.7] | 0 [0 to 0.7]
  Swelling: Any: number analyzed (Participants) | 564 | 562
  Swelling: Any | 9.2 [7.0 to 11.9] | 1.1 [0.4 to 2.3]
  Swelling: Mild: number analyzed (Participants) | 564 | 562
  Swelling: Mild | 6.2 [4.4 to 8.5] | 0.4 [0.0 to 1.3]
  Swelling: Moderate: number analyzed (Participants) | 564 | 562
  Swelling: Moderate | 3.0 [1.8 to 4.8] | 0.7 [0.2 to 1.8]
  Swelling: Severe: number analyzed (Participants) | 564 | 562
  Swelling: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Swelling: Grade 4: number analyzed (Participants) | 564 | 562
  Swelling: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Pain at the injection site: Any | 86.2 [83.0 to 88.9] | 13.9 [11.1 to 17.0]
  Pain at the injection site: Mild | 66.3 [62.2 to 70.2] | 13.5 [10.8 to 16.6]
  Pain at the injection site: Moderate | 19.9 [16.6 to 23.4] | 0.4 [0.0 to 1.3]
  Pain at the injection site: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Pain at the injection site: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions included redness, swelling, and pain at the injection site occurring at the BNT162b2 or placebo injection site. Local reactions were recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: greater than >2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, severe: >10.0 cm, and potentially life threatening (Grade 4): necrosis or exfoliative dermatitis. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity, and potentially life threatening (Grade 4): emergency room visit or hospitalization for severe pain. Exact 2-sided CI, based on the Clopper and Pearson method was used.
Time Frame: Within 7 Days After Vaccination 2
Population: Safety population included all participants who received any of the study intervention. Here, "Number of participants analyzed" included participants who received Vaccination 2 and signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 557 | 553
Percentage of participants
  Redness: Any | 0.2 [0.0 to 1.0] | 4.7 [3.1 to 6.8]
  Redness: Mild | 0.2 [0.0 to 1.0] | 4.3 [2.8 to 6.4]
  Redness: Moderate | 0 [0.0 to 0.7] | 0.4 [0.0 to 1.3]
  Redness: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Redness: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Swelling: Any | 0.4 [0.0 to 1.3] | 8.9 [6.6 to 11.5]
  Swelling: Mild | 0.4 [0.0 to 1.3] | 5.8 [4.0 to 8.1]
  Swelling: Moderate | 0 [0.0 to 0.7] | 3.1 [1.8 to 4.9]
  Swelling: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Swelling: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Pain at the injection site: Any | 6.6 [4.7 to 9.0] | 84.4 [81.2 to 87.4]
  Pain at the injection site: Mild | 6.3 [4.4 to 8.6] | 61.7 [57.5 to 65.7]
  Pain at the injection site: Moderate | 0.4 [0.0 to 1.3] | 22.4 [19.0 to 26.1]
  Pain at the injection site: Severe | 0 [0.0 to 0.7] | 0.4 [0.0 to 1.3]
  Pain at the injection site: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]

3. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events included fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain recorded by participants in an e-diary. Fever was defined as temperature: >=38.0 degrees (deg) Celsius (C), and categorized as: >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C, and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain, and new or worsened joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity, and severe: prevented daily routine activity. Vomiting graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h, severe: required intravenous hydration, and grade 4: emergency room (ER) visit or hospitalization for hypotensive shock. Diarrhea graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h, severe: 6 or more loose stools in 24h, and grade 4: ER visit or hospitalization for severe diarrhea.
Time Frame: Within 7 Days After Vaccination 1
Population: Safety population included all participants who received any of the study intervention. Here, "Number of participants analyzed" signifies number of participants evaluable and "Number Analyzed" (n) signifies number of participants evaluable for specified rows for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 564 | 563
Percentage of participants
  Fever: >=38.0 deg C: number analyzed (Participants) | 564 | 562
  Fever: >=38.0 deg C | 2.0 [1.0 to 3.5] | 1.1 [0.4 to 2.3]
  Fever: >=38.0 deg C to 38.4 deg C: number analyzed (Participants) | 564 | 562
  Fever: >=38.0 deg C to 38.4 deg C | 1.2 [0.5 to 2.5] | 0.4 [0.0 to 1.3]
  Fever: >38.4 deg C to 38.9 deg C: number analyzed (Participants) | 564 | 562
  Fever: >38.4 deg C to 38.9 deg C | 0.4 [0.0 to 1.3] | 0.4 [0.0 to 1.3]
  Fever: >38.9 deg C to 40.0 deg C: number analyzed (Participants) | 564 | 562
  Fever: >38.9 deg C to 40.0 deg C | 0.4 [0.0 to 1.3] | 0.4 [0.0 to 1.3]
  Fever: >40.0 deg C: number analyzed (Participants) | 564 | 562
  Fever: >40.0 deg C | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.7]
  Fatigue: Any | 64.0 [59.9 to 68.0] | 42.1 [38.0 to 46.3]
  Fatigue: Mild | 31.9 [28.1 to 35.9] | 24.7 [21.2 to 28.5]
  Fatigue: Moderate | 30.9 [27.1 to 34.8] | 16.3 [13.4 to 19.7]
  Fatigue: Severe | 1.2 [0.5 to 2.5] | 1.1 [0.4 to 2.3]
  Fatigue: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Headache: Any: number analyzed (Participants) | 564 | 562
  Headache: Any | 47.2 [43.0 to 51.4] | 34.3 [30.4 to 38.4]
  Headache: Mild: number analyzed (Participants) | 564 | 562
  Headache: Mild | 28.2 [24.5 to 32.1] | 23.3 [19.9 to 27.0]
  Headache: Moderate: number analyzed (Participants) | 564 | 562
  Headache: Moderate | 17.9 [14.8 to 21.3] | 10.3 [7.9 to 13.1]
  Headache: Severe: number analyzed (Participants) | 564 | 562
  Headache: Severe | 1.1 [0.4 to 2.3] | 0.7 [0.2 to 1.8]
  Headache: Grade 4: number analyzed (Participants) | 564 | 562
  Headache: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Chills: Any: number analyzed (Participants) | 564 | 562
  Chills: Any | 19.9 [16.6 to 23.4] | 6.2 [4.4 to 8.6]
  Chills: Mild: number analyzed (Participants) | 564 | 562
  Chills: Mild | 12.9 [10.3 to 16.0] | 4.3 [2.8 to 6.3]
  Chills: Moderate: number analyzed (Participants) | 564 | 562
  Chills: Moderate | 6.0 [4.2 to 8.3] | 1.6 [0.7 to 3.0]
  Chills: Severe: number analyzed (Participants) | 564 | 562
  Chills: Severe | 0.9 [0.3 to 2.1] | 0.4 [0.0 to 1.3]
  Chills: Grade 4: number analyzed (Participants) | 564 | 562
  Chills: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Vomiting: Any: number analyzed (Participants) | 564 | 562
  Vomiting: Any | 2.7 [1.5 to 4.3] | 0.9 [0.3 to 2.1]
  Vomiting: Mild: number analyzed (Participants) | 564 | 562
  Vomiting: Mild | 2.3 [1.2 to 3.9] | 0.7 [0.2 to 1.8]
  Vomiting: Moderate: number analyzed (Participants) | 564 | 562
  Vomiting: Moderate | 0.4 [0.0 to 1.3] | 0.2 [0.0 to 1.0]
  Vomiting: Severe: number analyzed (Participants) | 564 | 562
  Vomiting: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Vomiting: Grade 4: number analyzed (Participants) | 564 | 562
  Vomiting: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Diarrhea: Any: number analyzed (Participants) | 564 | 562
  Diarrhea: Any | 11.5 [9.0 to 14.5] | 10.1 [7.8 to 12.9]
  Diarrhea: Mild: number analyzed (Participants) | 564 | 562
  Diarrhea: Mild | 9.9 [7.6 to 12.7] | 8.9 [6.7 to 11.6]
  Diarrhea: Moderate: number analyzed (Participants) | 564 | 562
  Diarrhea: Moderate | 1.4 [0.6 to 2.8] | 1.2 [0.5 to 2.5]
  Diarrhea: Severe: number analyzed (Participants) | 564 | 562
  Diarrhea: Severe | 0.2 [0.0 to 1.0] | 0 [0.0 to 0.7]
  Diarrhea: Grade 4: number analyzed (Participants) | 564 | 562
  Diarrhea: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  New or worsened muscle pain: Any: number analyzed (Participants) | 564 | 562
  New or worsened muscle pain: Any | 27.7 [24.0 to 31.6] | 11.4 [8.9 to 14.3]
  New or worsened muscle pain: Mild: number analyzed (Participants) | 564 | 562
  New or worsened muscle pain: Mild | 15.8 [12.9 to 19.1] | 6.2 [4.4 to 8.6]
  New or worsened muscle pain: Moderate: number analyzed (Participants) | 564 | 562
  New or worsened muscle pain: Moderate | 11.3 [8.8 to 14.3] | 5.0 [3.3 to 7.1]
  New or worsened muscle pain: Severe: number analyzed (Participants) | 564 | 562
  New or worsened muscle pain: Severe | 0.5 [0.1 to 1.5] | 0.2 [0.0 to 1.0]
  New or worsened muscle pain: Grade 4: number analyzed (Participants) | 564 | 562
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  New or worsened joint pain: Any: number analyzed (Participants) | 564 | 562
  New or worsened joint pain: Any | 15.1 [12.2 to 18.3] | 5.3 [3.6 to 7.5]
  New or worsened joint pain: Mild: number analyzed (Participants) | 564 | 562
  New or worsened joint pain: Mild | 10.3 [7.9 to 13.1] | 2.7 [1.5 to 4.4]
  New or worsened joint pain: Moderate: number analyzed (Participants) | 564 | 562
  New or worsened joint pain: Moderate | 4.8 [3.2 to 6.9] | 2.7 [1.5 to 4.4]
  New or worsened joint pain: Severe: number analyzed (Participants) | 564 | 562
  New or worsened joint pain: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  New or worsened joint pain: Grade 4: number analyzed (Participants) | 564 | 562
  New or worsened joint pain: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]

4. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: Systemic events included fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain recorded by participants in an e-diary. Fever was defined as temperature: >=38.0 deg C, and categorized as: >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C, and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain, and new or worsened joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity, and severe: prevented daily routine activity. Vomiting graded as mild: 1 to 2 times in 24h, moderate: >2 times in 24h, severe: required intravenous hydration, and grade 4: ER visit or hospitalization for hypotensive shock. Diarrhea graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h, severe: 6 or more loose stools in 24h, and grade 4: ER visit or hospitalization for severe diarrhea. Exact 2-sided CI, based on Clopper and Pearson method used.
Time Frame: Within 7 Days After Vaccination 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 557 | 553
Percentage of participants
  Fever: >=38.0 deg C | 1.1 [0.4 to 2.3] | 1.6 [0.7 to 3.1]
  Fever: >=38.0 deg C to 38.4 deg C | 0.5 [0.1 to 1.6] | 1.1 [0.4 to 2.3]
  Fever: >38.4 deg C to 38.9 deg C | 0.5 [0.1 to 1.6] | 0.5 [0.1 to 1.6]
  Fever: >38.9 deg C to 40.0 deg C | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Fever: >40.0 deg C | 0. [0.0 to 0.7] | 0 [0.0 to 0.7]
  Fatigue: Any | 21.7 [18.4 to 25.4] | 50.8 [46.6 to 55.1]
  Fatigue: Mild | 12.4 [9.8 to 15.4] | 27.3 [23.6 to 31.2]
  Fatigue: Moderate | 8.6 [6.4 to 11.3] | 22.1 [18.7 to 25.8]
  Fatigue: Severe | 0.7 [0.2 to 1.8] | 1.4 [0.6 to 2.8]
  Fatigue: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Headache: Any | 20.8 [17.5 to 24.4] | 37.8 [33.7 to 42.0]
  Headache: Mild | 13.1 [10.4 to 16.2] | 25.0 [21.4 to 28.8]
  Headache: Moderate | 7.5 [5.5 to 10.1] | 12.1 [9.5 to 15.1]
  Headache: Severe | 0.2 [0.0 to 1.0] | 0.7 [0.2 to 1.8]
  Headache: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Chills: Any | 3.4 [2.1 to 5.3] | 13.4 [10.7 to 16.5]
  Chills: Mild | 2.3 [1.2 to 4.0] | 8.5 [6.3 to 11.1]
  Chills: Moderate | 1.1 [0.4 to 2.3] | 4.7 [3.1 to 6.8]
  Chills: Severe | 0 [0.0 to 0.7] | 0.2 [0.0 to 1.0]
  Chills: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Vomiting: Any | 1.1 [0.4 to 2.3] | 2.4 [1.3 to 4.0]
  Vomiting: Mild | 0.7 [0.2 to 1.8] | 1.8 [0.9 to 3.3]
  Vomiting: Moderate | 0.4 [0.0 to 1.3] | 0.5 [0.1 to 1.6]
  Vomiting: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Vomiting: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  Diarrhea: Any | 4.5 [2.9 to 6.6] | 6.5 [4.6 to 8.9]
  Diarrhea: Mild | 3.8 [2.3 to 5.7] | 5.2 [3.5 to 7.4]
  Diarrhea: Moderate | 0.7 [0.2 to 1.8] | 0.9 [0.3 to 2.1]
  Diarrhea: Severe | 0 [0.0 to 0.7] | 0.4 [0.0 to 1.3]
  Diarrhea: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  New or worsened muscle pain: Any | 5.2 [3.5 to 7.4] | 23.5 [20.0 to 27.3]
  New or worsened muscle pain: Mild | 2.7 [1.5 to 4.4] | 12.8 [10.2 to 15.9]
  New or worsened muscle pain: Moderate | 2.5 [1.4 to 4.2] | 10.5 [8.1 to 13.3]
  New or worsened muscle pain: Severe | 0 [0.0 to 0.7] | 0.2 [0.0 to 1.0]
  New or worsened muscle pain: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  New or worsened joint pain: Any | 3.4 [2.1 to 5.3] | 9.8 [7.4 to 12.5]
  New or worsened joint pain: Mild | 2.0 [1.0 to 3.5] | 5.6 [3.8 to 7.9]
  New or worsened joint pain: Moderate | 1.4 [0.6 to 2.8] | 4.2 [2.7 to 6.2]
  New or worsened joint pain: Severe | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]
  New or worsened joint pain: Grade 4 | 0 [0.0 to 0.7] | 0 [0.0 to 0.7]

5. Primary Outcome: Percentage of Participants With Adverse Events Within 1 Month After Vaccination 1
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided CI was calculated using the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Within 1 month after Vaccination 1
Population: Safety population included all participants who received any of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 564 | 564
Percentage of participants | 31.6 [27.7 to 35.6] | 30.5 [26.7 to 34.5]

6. Primary Outcome: Percentage of Participants With Adverse Events Within 1 Month After Vaccination 2
Description: as for outcome 5
Time Frame: Within 1 month after Vaccination 2
Population: Safety population included all participants who received any of the study intervention. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure''.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 562 | 557
Percentage of participants | 29.0 [25.3 to 32.9] | 25.1 [21.6 to 29.0]

7. Primary Outcome: Percentage of Participants With Serious Adverse Events Within 1 Month After Vaccination 1
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided CI was calculated using the Clopper and Pearson method. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; or that was considered to be an important medical event.
Time Frame: Within 1 Month After Vaccination 1
Population: Safety population included all participants who received any of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 564 | 564
Percentage of participants | 0.4 [0.0 to 1.3] | 0.2 [0.0 to 1.0]

8. Primary Outcome: Percentage of Participants With Serious Adverse Events Within 1 Month After Vaccination 2
Description: as for outcome 7
Time Frame: Within 1 Month After Vaccination 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 562 | 557
Percentage of participants | 0.5 [0.1 to 1.6] | 0.7 [0.2 to 1.8]

9. Primary Outcome: Geometric Mean Ratio (GMR) Based on Geometric Mean Concentration (GMC) of Full-Length S-binding Immunoglobulin G (IgG) at 1 Month After BNT162b2 Vaccination
Description: GMCs of full-length S-binding IgG level for the coadministration group and separate administration group were reported in this outcome measure in descriptive data section. GMC and the 2-sided 95% CI were calculated by exponentiating the LSMeans of the concentrations and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of vaccine group, age group, and the corresponding baseline assay results (log scale). Assay results below the LLOQ were set to 0.5*LLOQ. Geometric mean ratio (GMR) was reported in the statistical analysis section and was calculated as ratio of GMCs in the coadministration group to the separate administration group. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure.
Time Frame: 1 Month After BNT162b2 vaccination
Population: Evaluable BNT162b2 immunogenicity population: Eligible participants who received all vaccinations(Vax) at Visit1(V1) (coadministration group) or all Vax at V1 and V2 (separate administration group) as randomized, had at least 1 valid full-length S-binding IgG result from blood sample collected 28 to 42 days after BNT162b2 vax, had no reported COVID-19/new SARS-CoV-2 infection after V1 through 1 month after BNT162b2 vax, and had no other important protocol deviations as determined by clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Units per millilitre (U/mL)
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 499 | 413
Units per millilitre (U/mL) | 13767.8 [13110.0 to 14458.6] | 16644.5 [15774.7 to 17562.3]
Statistical Analysis 1: Comparison: Coadministration Group vs Separate Administration Group; Test type: Non-Inferiority — Noninferiority was declared if the lower bound of the 2-sided 95% CI for the GMR (coadministration group to separate-administration group) was greater than 0.67; GMR = 0.83, 95% CI 2-sided [0.77 to 0.89] — GMRs and 95% CIs were calculated by exponentiating LSmeans difference of logarithms of concentrations (coadmin group-separate admin group), corresponding CIs based on analysis of log transformed assay results using a linear regression model

10. Primary Outcome: Geometric Mean Ratio (GMR) Based on Geometric Mean Titer (GMT) of Strain-Specific Hemagglutination Inhibition (HAI) at 1 Month After SIIV Vaccination
Description: GMTs of strain-specific HAI titers for the coadministration group and separate administration group were reported in this outcome measure in descriptive data section. GMTs and the 2-sided 95% CIs were calculated by exponentiating the LSMeans of the titers and the corresponding CIs based on analysis of logarithmically transformed assay results using a linear regression model with terms of vaccine group, age group, and the corresponding baseline assay results (log scale). Assay results below the LLOQ were set to 0.5*LLOQ, and results above the ULOQ were set to ULOQ+1. Geometric mean ratio (GMR) was reported in the statistical analysis section and was calculated as ratio of GMT in the coadministration group to the separate administration group.
Time Frame: 1 Month After SIIV vaccination
Population: Evaluable SIIV immunogenicity population: participants who received all vaccinations at Visit 1 as randomized, had at least 1 valid and determinate HAI titer result from the blood sample collected 28 to 42 days after SIIV, and had no other important protocol deviations as determined by the clinician. Here, "Number of participants analyzed" signifies number of participants evaluable and "Number Analyzed" (n) signifies number of participants evaluable for specified rows for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 515 | 484
Titer
  B/Austria: number analyzed (Participants) | 511 | 480
  B/Austria | 80.1 [71.7 to 89.6] | 89.7 [80.0 to 100.7]
  B/Phuket | 81.3 [74.4 to 88.9] | 81.3 [74.2 to 89.2]
  H1N1 A/Victoria: number analyzed (Participants) | 508 | 478
  H1N1 A/Victoria | 301.7 [273.1 to 333.4] | 316.5 [285.5 to 350.9]
  H3N2 A/Darwin: number analyzed (Participants) | 514 | 482
  H3N2 A/Darwin | 226.8 [207.2 to 248.3] | 235.6 [214.6 to 258.7]
Statistical Analysis 1: Comparison: Coadministration Group vs Separate Administration Group; B/Austria; Test type: Non-Inferiority — Noninferiority was declared for an influenza strain if the lower bound of the 2-sided 95% CI for the GMR (coadministration group to separate administration group) was greater than 0.67; Geometric Mean Ratio = 0.89, 95% CI 2-sided [0.77 to 1.04] — GMRs and 95% CIs were calculated by exponentiating LSmeans difference of logarithms of titers (coadministration group-separate administration group), corresponding CIs based on analysis of log transformed assay results using a linear regression model
Statistical Analysis 2: Comparison: Coadministration Group vs Separate Administration Group; B/Phuket; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMR = 1.00, 95% CI 2-sided [0.89 to 1.13] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Coadministration Group vs Separate Administration Group; H1N1 A/Victoria; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMR = 0.95, 95% CI 2-sided [0.83 to 1.09] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Coadministration Group vs Separate Administration Group; H3N2 A/Darwin; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; GMR = 0.96, 95% CI 2-sided [0.85 to 1.09] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Geometric Mean Concentration (GMC) of Full-Length S-binding IgG Levels Before Vaccination and 1 Month After BNT162b2 Vaccination
Description: GMCs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student's t-distribution). Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLOQ. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure''.
Time Frame: Before BNT162b2 vaccination, and 1 month After BNT162b2 vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Units per millilitre (U/mL)
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 499 | 413
Units per millilitre (U/mL)
  Before BNT162b2 Vaccination | 5520.3 [5034.7 to 6052.8] | 5272.3 [4704.3 to 5909.0]
  1 Month After BNT162b2 Vaccination | 13806.5 [12838.9 to 14847.0] | 16254.6 [15035.5 to 17572.5]

12. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Full-Length S-binding IgG Levels From Before Vaccination to 1 Month After BNT162b2 Vaccination
Description: GMFR was defined as the geometric mean of the ratios of IgG concentrations at 1 month after BNT162b2 vaccination to that before BNT162b2 vaccination. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student's t-distribution). Assay results below the LLOQ were set to 0.5*LLOQ. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure''.
Time Frame: From before BNT162b2 vaccination to 1 month After BNT162b2 vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 499 | 413
Fold rise | 2.5 [2.4 to 2.7] | 3.1 [2.9 to 3.3]

13. Secondary Outcome: Geometric Mean Titer (GMT) of SARS-CoV-2 Neutralizing Titers Before Vaccination and 1 Month After BNT162b2 Vaccination
Description: GMTs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student's t-distribution). Assay results below LLOQ were set to 0.5*LLOQ. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure''. Analysis was performed in a subset of 100 participants from each group.
Time Frame: Before BNT162b2 vaccination, and 1 month after BNT162b2 vaccination
Population: Evaluable BNT162b2 immunogenicity population: Eligible participants who received all Vax at V1 (coadministration group) or all Vax at V1 and V2 (separate administration group) as randomized, had at least 1 valid SARS-CoV-2 neutralizing titers result from blood sample collected 28 to 42 days after BNT162b2 vax, had no reported COVID-19/new SARS-CoV-2 infection after V1 through 1 month after BNT162b2 vax, and had no other important protocol deviations as determined by clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 100 | 100
Titer
  Before BNT162b2 Vaccination | 2755.9 [2107.6 to 3603.4] | 2421.2 [1780.1 to 3293.3]
  1 Month After BNT162b2 Vaccination | 6773.9 [5545.0 to 8275.3] | 7886.6 [6264.9 to 9928.2]

14. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Neutralizing Titers From Before Vaccination to 1 Month After BNT162b2 Vaccination
Description: GMFR was defined as the geometric mean of the ratios of SARS-CoV-2 neutralizing titers at 1 month after BNT162b2 vaccination to that before BNT162b2 vaccination. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student's t-distribution). Assay results below the LLOQ were set to 0.5*LLOQ. Here, "Number of participants analyzed" signifies number of participants evaluable for this outcome measure''. Analysis was performed in a subset of 100 participants from each group.
Time Frame: From before BNT162b2 vaccination to 1 month after BNT162b2 vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 100 | 100
Fold rise | 2.5 [2.1 to 2.9] | 3.3 [2.7 to 3.9]

15. Secondary Outcome: Geometric Mean Titer (GMT) of Strain-Specific HAI Titers Before Vaccination and 1 Month After SIIV Vaccination
Description: GMTs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on the Student's t-distribution). Assay results below the LLOQ were set to 0.5*LLOQ, and results above the ULOQ were set to ULOQ+1. The analysis was performed on the influenza strains: H1N1 A/Victoria, H3N2 A/Darwin, B/Austria, and B/Phuket.
Time Frame: Before SIIV vaccination, and 1 month after SIIV vaccination
Population: Evaluable SIIV immunogenicity population: eligible randomized participants who received all vaccinations at Visit 1 as randomized, had at least 1 valid and determinate HAI titer result from the blood sample collected for 28 to 42 days after SIIV vax, and had no other important protocol deviations as determined by the clinician. Here, "N" signifies number of participants evaluable, and "n" signifies number of participants evaluable for specified rows for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 520 | 496
Titer
  B/Austria: Before Vaccination: number analyzed (Participants) | 515 | 483
  B/Austria: Before Vaccination | 13.0 [11.7 to 14.5] | 12.7 [11.5 to 14.1]
  B/Austria: 1 Month After SIIV Vaccination: number analyzed (Participants) | 514 | 491
  B/Austria: 1 Month After SIIV Vaccination | 72.4 [64.2 to 81.7] | 78.3 [69.3 to 88.5]
  B/Phuket: Before Vaccination: number analyzed (Participants) | 515 | 484
  B/Phuket: Before Vaccination | 26.4 [23.8 to 29.4] | 25.7 [23.0 to 28.6]
  B/Phuket: 1 Month After SIIV Vaccination | 87.4 [79.7 to 95.7] | 86.3 [78.4 to 94.9]
  H1N1 A/Victoria: Before Vaccination: number analyzed (Participants) | 509 | 478
  H1N1 A/Victoria: Before Vaccination | 57.0 [49.5 to 65.6] | 56.3 [48.9 to 64.7]
  H1N1 A/Victoria: 1 Month After SIIV Vaccination: number analyzed (Participants) | 516 | 492
  H1N1 A/Victoria: 1 Month After SIIV Vaccination | 344.3 [312.4 to 379.3] | 362.3 [326.8 to 401.6]
  H3N2 A/Darwin: Before Vaccination: number analyzed (Participants) | 514 | 482
  H3N2 A/Darwin: Before Vaccination | 39.5 [35.6 to 43.7] | 38.4 [34.5 to 42.8]
  H3N2 A/Darwin: 1 Month After SIIV Vaccination: number analyzed (Participants) | 519 | 491
  H3N2 A/Darwin: 1 Month After SIIV Vaccination | 230.6 [209.5 to 253.8] | 242.2 [221.2 to 265.2]

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Strain-Specific HAI Titers From Before Vaccination to 1 Month After SIIV Vaccination
Description: GMFR was defined as ratio of the geometric mean of strain-specific HAI titers at 1 month after SIIV vaccination to the geometric mean of strain-specific HAI titers before SIIV vaccination. GMFRs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student's t-distribution). Assay results below the LLOQ were set to 0.5*LLOQ, and results above the ULOQ were set to ULOQ+1. The analysis was performed on the influenza strains: H1N1 A/Victoria, H3N2 A/Darwin, B/Austria, and B/Phuket.
Time Frame: From before vaccination to 1 month after SIIV vaccination
Population: Evaluable SIIV immunogenicity population: eligible randomized participants who received all vaccinations at Visit 1 as randomized, had at least 1 valid and determinate HAI titer result from blood sample collected for 28 to 42 days after SIIV vax, and had no other important protocol deviations as determined by clinician. Here, "N" signifies number of participants evaluable, and "n" signifies number of participants evaluable for specified rows for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Coadministration Group | Separate Administration Group
Number analyzed (Participants) | 515 | 484
Fold rise
  B/Austria: number analyzed (Participants) | 511 | 480
  B/Austria | 5.5 [4.9 to 6.2] | 6.3 [5.6 to 7.1]
  B/Phuket | 3.3 [2.9 to 3.7] | 3.4 [3.0 to 3.8]
  H1N1 A/Victoria: number analyzed (Participants) | 508 | 478
  H1N1 A/Victoria | 6.0 [5.1 to 7.0] | 6.4 [5.5 to 7.5]
  H3N2 A/Darwin: number analyzed (Participants) | 514 | 482
  H3N2 A/Darwin | 5.9 [5.3 to 6.6] | 6.3 [5.6 to 7.1]

ADVERSE EVENTS:
Time Frame: AEs and SAEs: From Day 1 (Visit 1) to 1 month after last dose of study vaccine (approximately 2 months after Visit 1 [Day1]); Local reactions (at the BNT162b2/placebo injection site) and systemic events: Within 7 days after each vaccination
Description: An AE may be categorized as serious in 1 participant and non-serious in another participant, or 1 participant may experience both serious and non-serious AE during the study. Safety population included all participants who received any of the study intervention. AEs included events collected in electronic diary (local and systemic reactions; systematic assessment) and events collected on case report form at each visit (non-systematic assessment).
Groups:
- Coadministration Group (Visit 1); Coadministration Group (Visit 2): Participants were randomized to receive 30 microgram (mcg) intramuscular (IM) injection of BNT162b2 vaccine along with IM injection of Seasonal Inactivated Influenza Vaccine (SIIV) on Day 1 (Visit 1), and IM injection of Placebo 1 month later (Visit 2).
- Separate Administration Group (Visit 1); Separate Administration Group (Visit 2): Participants were randomized to receive an intramuscular (IM) injection of Placebo along with IM injection of Seasonal Inactivated Influenza Vaccine (SIIV) on Day 1 (Visit 1), and 30 mcg IM injection of BNT162b2 vaccine 1 month later (Visit 2).
Arm/Group | Coadministration Group (Visit 1) | Coadministration Group (Visit 2) | Separate Administration Group (Visit 1) | Separate Administration Group (Visit 2)
All-Cause Mortality (participants affected / at risk) | 0/564 | 0/562 | 0/564 | 0/557
Serious Adverse Events (participants affected / at risk) | 2/564 | 3/562 | 1/564 | 4/557
Other Adverse Events (participants affected / at risk) | 532/564 | 261/562 | 364/564 | 502/557
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coadministration Group (Visit 1) (N=564) | Coadministration Group (Visit 2) (N=562) | Separate Administration Group (Visit 1) (N=564) | Separate Administration Group (Visit 2) (N=557)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Coadministration Group (Visit 1) (N=564) | Coadministration Group (Visit 2) (N=562) | Separate Administration Group (Visit 1) (N=564) | Separate Administration Group (Visit 2) (N=557)
Diarrhoea (Gastrointestinal disorders) | 65 | 25 | 57 | 36
Vomiting (Gastrointestinal disorders) | 15 | 6 | 5 | 13
Chills (General disorders) | 112 | 19 | 35 | 74
Fatigue (General disorders) | 361 | 121 | 237 | 281
Influenza like illness (General disorders) | 9 | 9 | 12 | 7
Injection site erythema (General disorders) | 43 | 1 | 3 | 26
Injection site pain (General disorders) | 486 | 37 | 78 | 467
Injection site pain (General disorders) | 16 | 1 | 14 | 1
Injection site swelling (General disorders) | 52 | 2 | 6 | 49
Pyrexia (General disorders) | 11 | 6 | 6 | 9
COVID-19 (Infections and infestations) | 46 | 63 | 56 | 48
Gastroenteritis (Infections and infestations) | 8 | 6 | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 27 | 31 | 24 | 22
Viral upper respiratory tract infection (Infections and infestations) | 4 | 6 | 6 | 7
Headache (Nervous system disorders) | 266 | 116 | 193 | 209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT05310084/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05310084/SAP_001.pdf